CLINICAL TRIAL: NCT02716831
Title: Addressing Weight History to Improve Behavioral Treatments for Bulimia Nervosa
Brief Title: Improving Treatments for Bulimia Nervosa: Innovation in Psychological Interventions for Regulating Eating
Acronym: INSPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1501003366; 1K23MH105680-01A1 (NIH)
Record Dates: First submitted 2016-03-11; First posted 2016-03-23 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Bulimia Nervosa; Bulimia; Binge Eating; Purging (Eating Disorders); Eating Disorder
Keywords: Bulimia Nervosa; Eating Disorders; Binge Eating; Bulimia; Purging
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Feeding and Eating Disorders | interventions — Nutrition Assessment; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseling & Acceptance-based Therapy (Experimental): Nutritional Counseling & Acceptance-based Therapy (N-CAAT) incorporates acceptance-based behavioral strategies and nutritional counseling designed to encourage willingness to tolerate distress and the ability to pursue chosen values in an adaptive manner despite distressing internal experiences. In addition to these skills, a principal focus of the treatment will be on identifying, practicing, and achieving behavioral goals, such as normalization of eating, reduction of maladaptive dietary restraint and restriction, and elimination of compensatory behaviors.
  Interventions: Behavioral: Nutritional Counseling & Acceptance-based Therapy
- Cognitive Therapy for Eating Disorders (Active Comparator): Participants in the Cognitive Behavioral Therapy for Eating Disorders (CBT) condition will receive 20-sessions of standard CBT for eating disorders based on the treatment approach developed by Dr. Christopher Fairburn and published in his book Cognitive Behavioral Therapy and Eating Disorders.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Eating Disorders

INTERVENTIONS:
Behavioral: Nutritional Counseling & Acceptance-based Therapy
  Arms: Counseling & Acceptance-based Therapy
Behavioral: Cognitive Behavioral Therapy for Eating Disorders
  Arms: Cognitive Therapy for Eating Disorders

SUMMARY:
The purpose of the study is to test a novel, acceptance-based behavioral treatment for bulimia nervosa (BN) in adults. This treatment is a type of individual psychotherapy called Nutritional Counseling And Acceptance-Based Therapy (N-CAAT) that enhances existing cognitive behavioral therapy (CBT) for BN by incorporating acceptance-based behavioral strategies and nutritional counseling to help patients eliminate BN symptoms.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is an eating disorder characterized by a pattern of binge eating and compensatory behaviors as well as an overemphasis on body weight and shape in self-evaluation. BN has a lifetime prevalence rate of 1-3% and is associated with numerous psychiatric and medical complications. Cognitive behavioral therapy (CBT) is regarded as the gold-standard treatment for BN and the treatment approach with the most empirical support to date. However, although CBT has accumulated impressive empirical support for its effectiveness, CBT produces abstinence from binge eating and purging in only 30-50% of treatment completers. Furthermore, relapse is common and many individuals do not maintain treatment gains. Innovative treatments that can improve rates of remission among patients with BN and related disorders are sorely needed for bulimia nervosa and related eating disorders, particularly for individuals for whom existing treatments fail.

Existing CBT may be enhanced by incorporating acceptance-based behavioral strategies and nutritional counseling to help patients eliminate BN symptoms. Acceptance-based behavioral treatments (ABBTs) emphasize "changing what you can and accepting what you can't", which refers to a focus on learning how to accept and tolerate distressing internal experiences (e.g., thoughts, emotions, urges, physical sensations) that might not be directly under the patients' control while choosing to engage in adaptive behavioral choices that are within their control. Patients may benefit from the provision of more adaptive behavioral strategies to maintain weight in a healthy range, which is not a primary goal of existing behavioral treatments. Nutritional counseling (NC), which is designed to promote healthy, non-rigid dietary restraint and exercise habits, can lead to improvements in weight control that may also improve disordered eating behaviors. As described above, a primary maintenance factor for BN is the strict and rigid dieting behavior that triggers urges to binge. Several studies have indicated that the provision of healthy restraint strategies to patients with BN can reduce binge eating and purging behaviors, suggesting that this approach can be an effective treatment alone or in combination with other behavioral techniques.

Study Objectives-

* Test the feasibility, acceptability, and preliminary efficacy of Nutritional Counseling And Acceptance-based Therapy (N-CAAT) for bulimia nervosa (BN) in a small pilot RCT trial
* Assess the mechanisms of action to enhance treatment development
* Evaluate the feasibility of recruitment, randomization, retention, assessment procedures, and implementation of the novel treatment to enhance the probability of success in subsequent larger RCTs

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic Statistical Manual(DSM)-5 criteria for Bulimia Nervosa
* Age 18 or above

Exclusion Criteria:

* Body Mass Index (BMI) below 85% of ideal body weight or other medical complications that prevent ability to engage in outpatient treatment
* Acute suicide risk
* Co-morbid diagnosis of a psychotic disorder, bipolar disorder, or substance dependence
* Diagnosis of mental retardation or a pervasive development disorder
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Binge and purge frequency assessed by the Eating Disorder Examination (EDE) | Change from Baseline Binge and Purge Frequency at 5 months and 11 months
  Binge and purge frequency as assessed by the Eating Disorder Examination (EDE)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Change from Baseline BMI at 1 month, 3 months, 5 months, and 11 months
  Body Mass Index (BMI) will be assessed to ensure weight remains in a healthy range and to track weight change
Broader Psychological Functioning assessed by the Symptom Checklist-90-Revisited | Change from Baseline Symptom Checklist-90 Revisited at 1 month, 3 months, 5 months, and 11 months
  Broader psychological functioning will be assessed by the Symptom Checklist-90-Revisited (SC) which assesses a broad range of psychological problems and symptoms of psychopathology

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne S Juarascio, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Parker MN, Wilkinson ML, Hunt RA, Ortiz A, Manasse SM, Juarascio AS. Eating expectancies and hedonic hunger among individuals with bulimia-spectrum eating disorders who plan binge-eating episodes. Int J Eat Disord. 2022 Jan;55(1):120-124. doi: 10.1002/eat.23628. Epub 2021 Oct 13. PMID 34643949
- See also: For more information, please email edresearch@drexel.edu or call 215-553-7186 — http://drexel.edu/coas/academics/departments-centers/well-center/research/current-research-projects/